CLINICAL TRIAL: NCT00270205
Title: A Phase I/II, Randomized, Double-Blind Study to Evaluate the Safety, Tolerability, and Immunogenicity of LC002, a DermaVir Vaccine, in HIV-1-Infected Subjects Currently Under Treatment With Highly Active Antiretroviral Therapy (HAART)
Brief Title: Safety, Tolerability and Immune Response to LC002, an Experimental Therapeutic Vaccine, in Adults Receiving HAART
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A5176; 10126 (Registry Identifier: DAIDS ES); ACTG A5176
Record Dates: First submitted 2005-12-21; First posted 2005-12-26 (Estimated); Results first posted 2011-10-13 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2017-12

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections | interventions — LC-002; Vaccination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A: 0.1 mg DNA/participant vaccination at weeks 1,7,13 (Experimental): Participants receiving three separate low-dose vaccinations of LC002 (0.1 mg DNA/participant, 0.8 ml total, administered over two skin sites [on the left and right upper back] of 80 cm^2 each, 0.4 ml/site) at weeks 1, 7, and 13.
  Interventions: Biological: LC002 standard vaccination
- B (Experimental): Participants receiving three separate vaccinations of LC002 placebo (0.8 ml total, administered over two skin sites [on the left and right upper back] of 80 cm^2 each, 0.4 ml/site) at weeks 1, 7, and 13.
  Interventions: Biological: LC002 placebo vaccination
- C: 0.4 mg DNA/participant vaccination at weeks 1, 7, 13 (Experimental): Participants receiving three separate high-dose vaccinations of LC002 (0.4 mg DNA/participant, 3.2 ml total, administered over four skin sites [on the left and right upper back and left and right upper ventral thigh] of 80 cm^2 each, 0.8 ml/site) at weeks 1, 7, and 13.
  Interventions: Biological: LC002 high-dose vaccination
- D (Experimental): Participants receiving three separate vaccinations of LC002 placebo (3.2 ml total, administered over four skin sites [on the left and right upper back and left and right upper ventral thigh] of 80 cm^2 each, 0.8 ml/site) at weeks 1, 7, and 13.
  Interventions: Biological: LC002 placebo vaccination
- E: 0.4 mg DNA/participant vaccination at weeks 0,1,6,7,12,13 (Experimental): Participants receiving six separate high-dose vaccinations of LC002 (0.4 mg DNA/participant, 3.2 ml total, administered over four skin sites [on the left and right upper back and left and right upper ventral thigh] of 80 cm^2 each, 0.8 ml/site) at study entry and weeks 1, 6, 7, 12, and 13.
  Interventions: Biological: LC002 high-dose vaccination
- F (Experimental): Participants receiving six separate vaccinations of LC002 placebo (3.2 ml total, administered over four skin sites [on the left and right upper back and left and right upper ventral thigh] of 80 cm^2 each, 0.8 ml/site) at study entry and weeks 1, 6, 7, 12, and 13.
  Interventions: Biological: LC002 placebo vaccination

INTERVENTIONS:
Biological: LC002 standard vaccination — 0.1 mg DNA/participant, 0.8 ml total administered subcutaneously
  Arms: A: 0.1 mg DNA/participant vaccination at weeks 1,7,13
Biological: LC002 high-dose vaccination — 0.4 mg DNA/participant, 3.2 ml total administered subcutaneously
  Arms: C: 0.4 mg DNA/participant vaccination at weeks 1, 7, 13; E: 0.4 mg DNA/participant vaccination at weeks 0,1,6,7,12,13
Biological: LC002 placebo vaccination — Placebo vaccination administered subcutaneously
  Arms: B; D; F

SUMMARY:
LC002 is an experimental therapeutic vaccine designed to boost the immune response of people infected with HIV. The purpose of this study was to determine the safety and tolerability of and immune response to LC002 in HIV-1-infected adults who are currently receiving anti-HIV treatment.

DETAILED DESCRIPTION:
The use of highly active antiretroviral therapy (HAART) has dramatically improved the rates of survival, morbidity, and mortality among HIV-infected people throughout the world. However, the costs, long-term toxicity, and problems with adherence associated with HAART regimens make such treatment plans less than optimal for individuals seeking treatment for HIV infection. Also, because viral reservoirs cannot be eradicated, HIV-infected people must usually be on HAART indefinitely in order to keep their infection under control. While the mechanism is still unclear, the immune system weakens as HIV disease progresses. A therapeutic HIV vaccine given to HIV infected people may help to promote better immune responses. LC002 is a novel HIV therapeutic vaccine containing a DNA plasmid that codes for most of HIV-1's proteins. LC002 is a unique vaccine in that it is given through topical administration; this allows for Langerhans cells (immune cells located under the surface of the skin) to pick up the vaccine and deliver it to the lymph nodes, causing an immune reaction. This study evaluated the safety, tolerability, and immunogenicity of LC002 in HIV-infected adults currently receiving HAART.

There were three cohorts in this study which were enrolled sequentially. Participants in a given cohort were randomly assigned to receive either LC002 (6 participants) or placebo (2 participants).

* In Cohort 1, participants received three separate low-dose vaccinations of LC002 (Arm A: 0.1 mg DNA/participant, 0.8 ml total, administered over two skin sites of 80 cm^2 each, 0.4 ml/site) or 3 separate vaccinations of placebo (Arm B: 0.8 ml total, administered over two skin sites of 80 cm^2 each, 0.4 ml/site). Vaccinations were given over two skin sites on the left and right upper back. Participants received vaccinations at weeks 1, 7, and 13.
* In Cohort 2, participants received three separate high-dose vaccinations of LC002 (Arm C: 0.4 mg DNA/participant, 3.2 ml total, administered over four skin sites of 80 cm^2 each, 0.8 ml/site) or three separate vaccinations of placebo (Arm D: 3.2 ml total, administered over four skin sites of 80 cm^2 each, 0.8 ml/site). Vaccinations were given over four skin sites on the left and right upper back and left and right upper ventral thigh. Participants received vaccinations at weeks 1, 7, and 13.
* In Cohort 3, participants received six separate high-dose vaccinations of LC002 (Arm E: 0.4 mg DNA/participant, 3.2 ml total, administered over four skin sites of 80 cm^2 each, 0.8 ml/site) or six vaccinations of placebo (Arm F: 3.2 ml total, administered over four skin sites of 80 cm^2 each, 0.8 ml/site). Vaccinations were given over four skin sites on the left and right upper back and left and right upper ventral thigh. Participants received vaccinations at study entry and weeks 1, 6, 7, 12, and 13.

The decision to open the next cohort was made when all participants in the current cohort have remained on study for >=14 days after the second vaccination or prematurely discontinued from study or had a primary safety endpoint (see primary outcome measure definition). Dose escalation required no primary safety endpoint and on-study follow-up for >=6 participants in the previous cohort(s).

Prior to receiving the vaccine, the chosen vaccine administration site on the back or thigh was disinfected and exfoliated. A skin patch was applied to the site, and the vaccine solution was placed on the skin underneath the patch with a needleless syringe. Participants were allowed to remove the skin patch 3 hours post vaccination. For the first and second vaccinations, participants were required to remain at the clinic for 3 hours post-vaccination so study staff can assess for side effects. If no side effects occurred after the first two vaccinations, participants were required to stay at the clinic for only 30 minutes after receiving later vaccinations.

At the start of the study, participants were asked to keep a diary and record daily any side effects or skin irritation they may have experienced following vaccination. Participants were required to bring their diaries with them to their next clinic visit. Two days after vaccination, participants were followed-up by phone and were asked about any side effects they may have experienced. Participants who experienced side effects were asked to return to the clinic for examination. There were 13 study visits; they occurred at study entry and Weeks 1, 3, 6, 7, 9, 12, 13, 15, 17, 24, 37, and 61. Study visits included medication history, a physical exam, and collection of diaries. Blood and urine collection occurred at selected visits. HAART was not be provided by the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-infected
* On a stable HAART regimen without changes or interruptions for more than 4 consecutive days for at least 12 weeks prior to study entry. Patients must be currently taking regimens containing drugs of at least two different classes.
* Two readings of plasma HIV-1 viral load of less than 50 copies/ml within 30 days prior to study entry. More information on this criterion can be found in the protocol.
* CD4 count greater than 350 cells/mm^3 within 12 weeks prior to study entry
* Lowest CD4 count greater than 250 cells/mm^3 at any time prior to study entry
* Willing to use acceptable forms of contraception
* Karnofsky performance score 90 or higher obtained within 30 days prior to study entry

Exclusion Criteria:

* HIV-1 viral load greater than 500 copies/ml within the 24 weeks prior to study entry
* History of or current active skin disease (e.g., atopic dermatitis, psoriasis) or any chronic autoimmune disease (e.g., Graves' disease). Participants with minor, localized skin conditions that, in the opinion of the investigator, do not represent a safety concern, are not excluded.
* Treatment with topical corticosteroids at the proposed vaccination sites (Cohort 1: left and right upper back; Cohorts 2 and 3: left and right upper back and left and right upper ventral thigh) within 2 weeks of study entry
* Excessive exposure to the sun (e.g., sunbathing, tanning bed) within 2 weeks prior to study entry
* Laser hair removal within 2 weeks prior to study entry
* Use of any local skin treatments (e.g., topical/chemical hair removal, ointments, possible irritants) to the targeted vaccination sites within 7 days prior to study entry
* History of diabetes or bleeding disorders
* Previous CDC Category C event. More information on this criterion can be found in the protocol.
* Use of immunomodulating therapy, including cyclosporine, IgG-containing products, interleukins, interferons, or systemic glucocorticosteroids (including those inhaled) within 6 months prior to study entry
* Exposure to an experimental HIV vaccine within 6 months prior to study entry
* Any vaccine within 30 days prior to study entry
* Investigational products within 12 weeks prior to study entry
* Allergy or sensitivity to study vaccine products, adhesives, or polyester
* Current drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with the study
* Serious illness requiring systemic treatment and/or hospitalization. Participants who complete therapy or are clinically stable on therapy for at least 14 days prior to study entry are not excluded.
* Positive hepatitis B surface antigen or positive anti-hepatitis C antibody at screening
* History of treatment with HAART during primary infection
* History of lymph node irradiation
* Pregnant or breastfeeding
* Certain abnormal laboratory results. More information on this criterion can be found in the protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2006-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benigno Rodriguez, MD, Study Chair — Division of Infectious Diseases ACTU, University Hospital of Cleveland, Cleveland, OH, USA
Locations (5):
- United States (5):
  - Univ. of California Davis Med. Ctr., ACTU, Sacramento, California
  - Chicago Children's CRS, Chicago, Illinois
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Lisziewicz J, Trocio J, Xu J, Whitman L, Ryder A, Bakare N, Lewis MG, Wagner W, Pistorio A, Arya S, Lori F. Control of viral rebound through therapeutic immunization with DermaVir. AIDS. 2005 Jan 3;19(1):35-43. doi: 10.1097/00002030-200501030-00004. PMID 15627031
- [Background] Lori F, Trocio J, Bakare N, Kelly LM, Lisziewicz J. DermaVir, a novel HIV immunisation technology. Vaccine. 2005 Mar 18;23(17-18):2030-4. doi: 10.1016/j.vaccine.2005.01.004. PMID 15755566
- [Background] Lori F, Weiner DB, Calarota SA, Kelly LM, Lisziewicz J. Cytokine-adjuvanted HIV-DNA vaccination strategies. Springer Semin Immunopathol. 2006 Nov;28(3):231-8. doi: 10.1007/s00281-006-0047-y. Epub 2006 Oct 20. PMID 17053912
- [Background] Rajcani J, Mosko T, Rezuchova I. Current developments in viral DNA vaccines: shall they solve the unsolved? Rev Med Virol. 2005 Sep-Oct;15(5):303-25. doi: 10.1002/rmv.467. PMID 15906276
- [Background] Somogyi E, Xu J, Gudics A, Toth J, Kovacs AL, Lori F, Lisziewicz J. A plasmid DNA immunogen expressing fifteen protein antigens and complex virus-like particles (VLP+) mimicking naturally occurring HIV. Vaccine. 2011 Jan 17;29(4):744-53. doi: 10.1016/j.vaccine.2010.11.019. Epub 2010 Nov 23. PMID 21109034
- [Background] Lorincz O, Toke ER, Somogyi E, Horkay F, Chandran PL, Douglas JF, Szebeni J, Lisziewicz J. Structure and biological activity of pathogen-like synthetic nanomedicines. Nanomedicine. 2012 May;8(4):497-506. doi: 10.1016/j.nano.2011.07.013. Epub 2011 Aug 10. PMID 21839051
- [Background] Toke ER, Lorincz O, Somogyi E, Lisziewicz J. Rational development of a stable liquid formulation for nanomedicine products. Int J Pharm. 2010 Jun 15;392(1-2):261-7. doi: 10.1016/j.ijpharm.2010.03.048. Epub 2010 Mar 25. PMID 20347027
- [Background] Cristillo AD, Lisziewicz J, He L, Lori F, Galmin L, Trocio JN, Unangst T, Whitman L, Hudacik L, Bakare N, Whitney S, Restrepo S, Suschak J, Ferrari MG, Chung HK, Kalyanaraman VS, Markham P, Pal R. HIV-1 prophylactic vaccine comprised of topical DermaVir prime and protein boost elicits cellular immune responses and controls pathogenic R5 SHIV162P3. Virology. 2007 Sep 15;366(1):197-211. doi: 10.1016/j.virol.2007.04.012. Epub 2007 May 11. PMID 17499328
- [Background] Lisziewicz J, Trocio J, Whitman L, Varga G, Xu J, Bakare N, Erbacher P, Fox C, Woodward R, Markham P, Arya S, Behr JP, Lori F. DermaVir: a novel topical vaccine for HIV/AIDS. J Invest Dermatol. 2005 Jan;124(1):160-9. doi: 10.1111/j.0022-202X.2004.23535.x. PMID 15654970
- [Background] Lisziewicz J, Rosenberg E, Lieberman J, Jessen H, Lopalco L, Siliciano R, Walker B, Lori F. Control of HIV despite the discontinuation of antiretroviral therapy. N Engl J Med. 1999 May 27;340(21):1683-4. doi: 10.1056/NEJM199905273402114. No abstract available. PMID 10348681
- [Background] Calarota SA, Foli A, Maserati R, Baldanti F, Paolucci S, Young MA, Tsoukas CM, Lisziewicz J, Lori F. HIV-1-specific T cell precursors with high proliferative capacity correlate with low viremia and high CD4 counts in untreated individuals. J Immunol. 2008 May 1;180(9):5907-15. doi: 10.4049/jimmunol.180.9.5907. PMID 18424710
- [Background] Gudmundsdotter L, Wahren B, Haller BK, Boberg A, Edback U, Bernasconi D, Butto S, Gaines H, Imami N, Gotch F, Lori F, Lisziewicz J, Sandstrom E, Hejdeman B. Amplified antigen-specific immune responses in HIV-1 infected individuals in a double blind DNA immunization and therapy interruption trial. Vaccine. 2011 Jul 26;29(33):5558-66. doi: 10.1016/j.vaccine.2011.01.064. Epub 2011 Feb 5. PMID 21300092
- [Result] Natz E, Lisziewicz J. Rational Design of Formulated DNA Vaccines: The DermaVir Approach. In J. Thalhamer, R. Weiss & S. Scheiblhofer (Eds.), Gene Vaccines. In press.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from February 2006 to October 2008 in 5 different U.S. sites. Enrollment was done by cohort with each cohort enrolling six participants for LC002 vaccine and 2 participants for its corresponding placebo. Cohorts were enrolled sequentially, with later cohorts receiving higher dose of the LC002 vaccine.
Pre-assignment Details: Study participants were HIV-1-infected men and women 18-50 years of age with CD4 count >350 cells/mm^3 and plasma HIV-1 RNA <50 copies/ml (on an ultrasensitive assay) and who were on a stable HAART regimen. One enrolled participant never started study treatment/vaccination.
Groups:
- A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13: Participants receiving three separate low-dose vaccinations of LC002 (0.1 mg DNA/participant, 0.8 ml total, administered over two skin sites [on the left and right upper back] of 80 cm^2 each, 0.4 ml/site) at weeks 1, 7, and 13.
- Placebo: All participants receiving vaccinations of LC002 placebo were combined together in this arm/group. This includes those participants in arms B, D and F.
Period: Overall Study
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Started | 6 | 6 (7 participants enrolled. One never started study vaccination and was excluded from all analyses.) | 6 | 7
Completed | 5 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age (in years) at study entry. Participants who never started study vaccination were excluded.
  years | 44 [32 to 48] | 41 [38 to 43] | 46 [34 to 47] | 34 [30 to 35] | 39 [32 to 45]
Age, Customized [Number; unit: participants] — Age (in years) at study entry. Participants who never started study vaccination were excluded.
  participants
    18-30 | 1 | 1 | 1 | 2 | 5
    31-40 | 2 | 2 | 1 | 5 | 10
    41-50 | 3 | 3 | 4 | 0 | 10
Sex: Female, Male [Count of Participants; unit: Participants] — Participants who never started study vaccination were excluded.
  Participants
    Female | 1 | 0 | 0 | 1 | 2
    Male | 5 | 6 | 6 | 6 | 23
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Primary Safety Endpoint
Description: Primary safety endpoint is defined as occurrence of at least one grade 3 or higher adverse event, including signs/symptoms, lab toxicities, and/or clinical events that is possibly or definitely related to study treatment. Event's relationship to the study treatment was determined by the protocol core team, including site clinicians on the team, blinded to the treatment arm. Adverse events solely attributed to an allergic reaction to the adhesive of the tape used to adhere the vaccination patch to the skin and not the vaccine itself were not used in determination of the primary safety endpoint.
Time Frame: From start of study vaccination to 28 days after the last study vaccination
Population: Only those participants who started study treatment/vaccination were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7
percentage of participants | 0 [0 to 40.2] | 0 [0 to 40.2] | 0 [0 to 40.2] | 0 [0 to 37.7]

2. Secondary Outcome: Time-averaged Area Under the Curve (AUC) of CD4+ T-cell Count in PBMCs
Description: Area under the curve (AUC) using linear trapezoidal method, of CD4+ T-cell count responses was used to characterize each participant's overall CD4+ count response. Each AUC was divided by 61 weeks to have the same unit as the raw data.
Time Frame: From start of study vaccination to week 61
Population: Only those participants who started study vaccination and who have complete and non-missing CD4+ T-cell count responses at all study visits were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 4 | 5 | 5
cells/mm3 | 735.0 [658.0 to 765.0] | 1169.5 [752.0 to 1424.5] | 745.0 [484.0 to 765.0] | 731.0 [552.0 to 769.0]

3. Secondary Outcome: Time-averaged AUC of CD8+ T-cell Count in PBMCs
Description: Area under the curve (AUC) using linear trapezoidal method, of CD8+ T-cell count responses was used to characterize each participant's overall CD8+ count response. Each AUC was divided by 61 weeks to have the same unit as the raw data.
Time Frame: From start of study vaccination to week 61
Population: Only those participants who started study vaccination and who have complete and non-missing CD8+ T-cell count responses at all study visits were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 4 | 5 | 5
cells/mm^3 | 612.0 [601.0 to 682.0] | 1061.0 [539.0 to 1402.0] | 686.0 [590.0 to 697.0] | 587.0 [483.0 to 842.0]

4. Secondary Outcome: Time-averaged AUC of the Magnitude of HIV-specific Immune Response, as Determined by Taking the Mean of the Number of Spot-forming Cells/10^6 PBMCs Observed in Each PHPC Assay for IFN-gamma Production for Gag p17, Gag p24, Gag p15 and Tat/Rev.
Description: At each week, the mean spot-forming cells/10^6 PBMCs detected by the PHPC (precursors with high proliferative capacity) assay across gag p17, gag p24, gag p15 and tat/rev was obtained per participant. Area under the curve (AUC) using linear trapezoidal method was used to characterize each participant's overall response. Each AUC was divided by 37 weeks to have the same unit of measure as the raw data.
Time Frame: From start of study vaccination to week 37
Population: Only those participants who started study vaccination and who have complete and non-missing mean responses to gag-1, gag-2, gag-3 and tat/rev through 37 weeks were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: spot-forming cells/10^6 PBMC
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 6
spot-forming cells/10^6 PBMC | 16441.8 [1896.1 to 37519.0] | 25797.0 [4708.3 to 46438.4] | 920.1 [133.6 to 4817.9] | 1760.4 [650.0 to 3122.9]

5. Secondary Outcome: Time-averaged AUC of the Magnitude of HIV-specific Immune Response, as Determined by the Number of Spot-forming Cells/10^6 PBMCs Observed in Each PHPC Assay for IFN-gamma Production for Gag p17, Gag p24, Gag p15 and Tat/Rev.
Description: Area under the curve (AUC) using linear trapezoidal method for each antigen was used to characterize each participant's overall response to the antigen as detected by the PHPC assay. Each AUC was divided by 37 weeks to have the same unit of measure as the raw data.
Time Frame: From start of study vaccination to week 37
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: spot-forming cells/10^6 PBMC
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 6
spot-forming cells/10^6 PBMC
  gag p17 | 18779.2 [2232.8 to 25283.1] | 6653.5 [4282.8 to 7466.4] | 1422.0 [104.5 to 7798.8] | 3120.7 [1076.0 to 6756.2]
  gag p24 | 15691.4 [2351.1 to 89228.3] | 33446.0 [6903.0 to 77524.8] | 585.1 [244.8 to 1360.1] | 641.2 [292.7 to 1749.9]
  gag p15 | 17977.7 [723.8 to 23520.9] | 13921.4 [6206.1 to 60107.5] | 1163.5 [163.9 to 2340.1] | 2244.4 [91.5 to 3349.3]
  tat/rev | 1272.0 [630.2 to 5226.8] | 2912.0 [2168.3 to 9518.1] | 268.3 [38.8 to 1149.9] | 712.8 [18.8 to 2035.2]

6. Secondary Outcome: Time-averaged AUC of the Magnitude of HIV-specific Immune Response, as Determined by Taking the Mean of the Number of Spot-forming Cells/10^6 PBMCs Observed in Each ELISPOT Assay for IFN-gamma Production for Gag p17, Gag p24, Gag p15 and Tat/Rev.
Description: At each week, the mean spot-forming cells/10^6 PBMCs across gag p17, gag p24, gag 15 and tat/rev was obtained per participant. Area under the curve (AUC) using linear trapezoidal method was used to characterize each participant's overall response. Each AUC was divided by 37 weeks to have the same unit of measure as the raw data.
Time Frame: From start of study vaccination to week 37
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: spot-forming cells/10^6 PBMC
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6
spot-forming cells/10^6 PBMC | 421.8 [401.8 to 443.0] | 274.5 [134.0 to 784.1] | 214.2 [59.4 to 576.2] | 126.7 [68.7 to 145.3]

7. Secondary Outcome: Time-averaged AUC of the Magnitude of HIV-specific Immune Response, as Determined by the Number of Spot-forming Cells/10^6 PBMCs Observed in Each ELISPOT Assay for IFN-gamma Production for Gag p17, Gag p24, Gag p15 and Tat/Rev.
Description: Area under the curve (AUC) using linear trapezoidal method for each antigen was used to characterize each participant's overall response to the antigen. Each AUC was divided by 37 weeks to have the same unit of measure as the raw data.
Time Frame: From start of study vaccination to week 37
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: spot-forming cells/10^6 PBMC
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6
spot-forming cells/10^6 PBMC
  gag p17 | 270.9 [130.0 to 364.7] | 186.5 [25.8 to 332.5] | 409.8 [159.8 to 1028.9] | 152.6 [57.8 to 234.1]
  gag p24 | 213.6 [113.0 to 795.9] | 458.4 [345.6 to 1999.4] | 135.3 [54.3 to 1193.5] | 103.8 [29.1 to 256.9]
  gag p15 | 141.5 [85.4 to 379.5] | 345.8 [31.5 to 386.1] | 31.0 [14.4 to 184.6] | 95.4 [35.0 to 277.5]
  tat/rev | 7.9 [6.0 to 419.6] | 22.9 [5.9 to 174.6] | 31.7 [15.3 to 133.5] | 33.3 [7.0 to 55.3]

8. Secondary Outcome: Anti-dsDNA Antibody Response
Description: Results report the number of participants who had negative anti-dsDNA antibody result at baseline and at week 17 or 61.
Time Frame: From start of study vaccination to week 61
Population: All participants who started study vaccination and who have anti-ds DNA results at baseline and week 17 or 61 were included in the analysis.
Measure: Number; unit: participants
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6
participants | 5 | 6 | 6 | 6

9. Secondary Outcome: Time-averaged AUC of T-cell Count of HIV-1-specific CD4+ T-cell Subsets, Based on Flow Cytometry With CFSE Staining to Detect Antigen-specific Lymphocyte Proliferation Responding to p24 Protein, Gag/Pol/Env and Tat/Rev
Description: Area under the curve (AUC) using linear trapezoidal method was used to characterize each participant's overall response. Each AUC was divided by 24 weeks to have the same unit of measure as the raw data.
Time Frame: From start of study vaccination to week 24
Population: Only those participants who started study vaccination and who have complete and non-missing responses through 24 weeks were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 6
cells/mm3
  p24 | 46.4 [44.8 to 91.7] | 21.5 [11.4 to 26.7] | 27.1 [13.2 to 32.3] | 13.0 [5.1 to 19.3]
  gag/pol/env | 27.5 [12.5 to 36.7] | 9.2 [8.0 to 20.5] | 8.4 [7.8 to 22.2] | 16.8 [0.5 to 25.7]
  tat/rev | 4.0 [1.1 to 14.2] | 4.0 [1.2 to 8.6] | 0.2 [0 to 0.3] | 10.1 [1.8 to 14.7]

10. Secondary Outcome: Time-averaged AUC of T-cell Count of HIV-1-specific CD4+ T-cell Subsets, Based on Flow Cytometry With CFSE Staining to Detect Antigen-specific Lymphocyte Proliferation Responding to Whole HIV-1 Antigen
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: Only those participants who started study vaccination and who have complete and non-missing responses through 24 weeks to whole HIV-1 antigen were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 3 | 6
cells/mm^3 | 305.3 [19.5 to 328.3] | 68.6 [6.2 to 459.0] | 4.6 [0 to 28.9] | 6.0 [3.5 to 73.0]

11. Secondary Outcome: Time-averaged AUC of T-cell Count of HIV-1-specific CD4+ T-cell Subsets, Based on Flow Cytometry With CFSE Staining to Detect Antigen-specific Lymphocyte Proliferation Responding to Anti-CD3
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: Only those participants who started study vaccination and who have complete and non-missing responses through 24 weeks to anti-CD3 antigen were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 5
cells/mm^3 | 333.6 [298.5 to 355.4] | 334.9 [210.4 to 548.6] | 200.4 [182.0 to 274.2] | 248.8 [213.4 to 293.3]

12. Secondary Outcome: Time-averaged AUC of T-cell Percent of HIV-1-specific CD4+ T-cell Subsets, Based on Flow Cytometry With CFSE Staining to Detect Antigen-specific Lymphocyte Proliferation Responding to p24 Protein, Gag/Pol/Env and Tat/Rev.
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 6
percent
  p24 | 10.0 [6.7 to 11.3] | 3.5 [1.2 to 4.6] | 4.9 [1.4 to 6.9] | 2.0 [0.7 to 3.1]
  gag/pol/env | 4.3 [1.7 to 4.7] | 1.4 [1.1 to 2.2] | 1.8 [0.9 to 2.2] | 2.5 [0.1 to 3.7]
  tat/rev | 0.6 [0.2 to 1.7] | 0.3 [0.1 to 1.9] | 0 [0 to 0.1] | 1.4 [0.2 to 1.8]

13. Secondary Outcome: Time-averaged AUC of T-cell Percent of HIV-1-specific CD4+ T-cell Subsets, Based on Flow Cytometry With CFSE Staining to Detect Antigen-specific Lymphocyte Proliferation Responding to Whole HIV-1 Antigen
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 3 | 6
percent | 42.0 [3.0 to 64.8] | 10.6 [1.7 to 44.2] | 1.1 [0 to 7.1] | 0.9 [0.5 to 15.2]

14. Secondary Outcome: Time-averaged AUC of T-cell Percent of HIV-1-specific CD4+ T-cell Subsets, Based on Flow Cytometry With CFSE Staining to Detect Antigen-specific Lymphocyte Proliferation Responding to Anti-CD3
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 5
percent | 47.7 [41.3 to 51.8] | 37.4 [35.7 to 53.7] | 31.1 [31.1 to 38.3] | 48.5 [36.2 to 49.1]

15. Secondary Outcome: Time-averaged AUC of T-cell Count of HIV-1-specific CD8+ T-cell Subsets, Based on Flow Cytometry With CFSE Staining to Detect Antigen-specific Lymphocyte Proliferation Responding to p24 Protein, Gag/Pol/Env, Tat/Rev and Whole HIV-1 Antigen.
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: Only those participants who started study vaccination and who have complete and non-missing responses through week 24 were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 6
cells/mm^3
  p24 | 10.5 [5.3 to 14.7] | 11.1 [3.5 to 12.0] | 1.0 [0.8 to 5.0] | 2.5 [0.8 to 5.1]
  gag/pol/env | 88.7 [72.8 to 107.0] | 59.1 [34.4 to 68.4] | 38.2 [22.4 to 62.2] | 44.3 [31.6 to 49.4]
  tat/rev | 2.5 [2.2 to 45.5] | 4.8 [1.7 to 17.1] | 5.7 [0.2 to 17.4] | 3.8 [1.6 to 6.1]
  HIV-1 MN | 118.6 [43.9 to 169.0] | 120.3 [60.9 to 130.9] | 73.5 [53.3 to 111.9] | 89.7 [37.1 to 118.5]

16. Secondary Outcome: Time-averaged AUC of T-cell Count of HIV-1-specific CD8+ T-cell Subsets, Based on Flow Cytometry With CFSE Staining to Detect Antigen-specific Lymphocyte Proliferation Responding to Anti-CD3
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5
cells/mm^3 | 330.6 [313.7 to 331.1] | 486.2 [458.6 to 727.9] | 350.4 [332.3 to 375.6] | 278.9 [222.2 to 449.4]

17. Secondary Outcome: Time-averaged AUC of T-cell Percent of HIV-1-specific CD8+ T-cell Subsets, Based on Flow Cytometry With CFSE Staining to Detect Antigen-specific Lymphocyte Proliferation Responding to p24 Protein, Gag/Pol/Env, Tat/Rev and Whole HIV-1 Antigen.
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 6
percent
  p24 | 2.1 [1.0 to 2.6] | 0.7 [0.4 to 1.4] | 0.1 [0.1 to 0.6] | 0.5 [0.1 to 0.7]
  gag/pol/env | 14.3 [9.9 to 15.1] | 4.8 [1.5 to 7.4] | 6.0 [3.0 to 7.4] | 6.0 [5.2 to 11.7]
  tat/rev | 0.5 [0.3 to 4.0] | 0.4 [0.2 to 1.0] | 1.1 [0 to 2.6] | 0.5 [0.3 to 0.7]
  HIV-1 MN | 24.9 [7.5 to 26.0] | 7.5 [6.1 to 12.0] | 10.4 [7.0 to 16.5] | 15.4 [6.5 to 16.7]

18. Secondary Outcome: Time-averaged AUC of T-cell Percent of HIV-1-specific CD8+ T-cell Subsets, Based on Flow Cytometry With CFSE Staining to Detect Antigen-specific Lymphocyte Proliferation Responding to Anti-CD3
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 5
percent | 58.4 [57.5 to 62.7] | 54.3 [34.5 to 67.7] | 48.5 [43.2 to 63.9] | 53.5 [47.9 to 62.5]

19. Secondary Outcome: Time-averaged AUC of T-cell Count of HIV-1-specific CD4+ T-cell Subsets, Based on Flow Cytometry to Detect Antigen-specific IFN-gamma-producing Cells Responding to Whole Zn-finger Inactivated Virus Stimulation and Various HIV-1 Peptide Antigens
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 4 | 6
cells/mm^3
  HIV-1 MN | 1.2 [0.7 to 1.4] | 0.3 [0 to 0.5] | 0.1 [0 to 0.3] | 0 [0 to 0]
  gag/pol/env | 0.7 [0.7 to 1.0] | 0 [0 to 0.1] | 0.1 [0 to 0.3] | 0 [0 to 0.2]
  tat/rev | 0.4 [0.3 to 0.8] | 0.3 [0.2 to 0.3] | 0 [0 to 0] | 0.2 [0 to 0.6]
  SEB | 18.3 [17.4 to 21.7] | 24.2 [7.6 to 65.4] | 6.1 [4.7 to 23.5] | 10.4 [7.4 to 18.4]

20. Secondary Outcome: Time-averaged AUC of T-cell Percent of HIV-1-specific CD4+ T-cell Subsets, Based on Flow Cytometry to Detect Antigen-specific IFN-gamma-producing Cells Responding to Whole Zn-finger Inactivated Virus Stimulation and Various HIV-1 Peptide Antigens
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 4 | 6
percent
  HIV-1 MN | 0.2 [0.1 to 0.2] | 0 [0 to 0.1] | 0 [0 to 0.1] | 0 [0 to 0]
  gag/pol/env | 0.1 [0.1 to 0.2] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0.1]
  tat/rev | 0.1 [0 to 0.1] | 0 [0 to 0.1] | 0 [0 to 0] | 0 [0 to 0.1]
  SEB | 2.6 [2.2 to 2.9] | 3.6 [1.1 to 8.2] | 1.2 [1.0 to 3.7] | 2.0 [1.4 to 2.4]

21. Secondary Outcome: Time-averaged AUC of T-cell Count of HIV-1-specific CD8+ T-cell Subsets, Based on Flow Cytometry to Detect Antigen-specific IFN-gamma-producing Cells Responding to Whole Zn-finger Inactivated Virus Stimulation and Various HIV-1 Peptide Antigens
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 5 | 4 | 6
cells/mm^3
  HIV-1 MN | 0.4 [0 to 0.4] | 0.3 [0.2 to 0.5] | 0 [0 to 0.5] | 0 [0 to 0.1]
  gag/pol/env | 3.1 [1.0 to 3.2] | 2.0 [1.9 to 10.5] | 1.0 [0.2 to 1.8] | 1.0 [0.1 to 2.0]
  tat/rev | 2.2 [0.4 to 5.6] | 0.5 [0.5 to 1.2] | 0.3 [0.1 to 0.7] | 1.1 [0.6 to 1.9]
  SEB | 19.2 [11.0 to 25.5] | 31.4 [25.0 to 35.9] | 32.2 [16.2 to 49.1] | 17.2 [9.4 to 30.6]

22. Secondary Outcome: Time-averaged AUC of T-cell Percent of HIV-1-specific CD8+ T-cell Subsets, Based on Flow Cytometry to Detect Antigen-specific IFN-gamma-producing Cells Responding to Whole Zn-finger Inactivated Virus Stimulation and Various HIV-1 Peptide Antigens
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 4 | 6
percent
  HIV-1 MN | 0 [0 to 0.1] | 0 [0 to 0.1] | 0 [0 to 0.1] | 0 [0 to 0]
  gag/pol/env | 0.5 [0.1 to 0.7] | 0.2 [0.2 to 0.6] | 0.2 [0.1 to 0.3] | 0.1 [0 to 0.3]
  tat/rev | 0.3 [0.1 to 0.9] | 0.1 [0 to 0.3] | 0.1 [0 to 0.1] | 0.2 [0.1 to 0.3]
  SEB | 4.0 [3.0 to 4.1] | 4.9 [1.7 to 6.0] | 5.1 [3.7 to 6.8] | 3.1 [2.8 to 3.3]

23. Secondary Outcome: Time-averaged AUC of T-cell Count of HIV-1-specific CD4+ T-cell Subsets, Based on Flow Cytometry to Detect Antigen-specific IL-2-producing Cells Responding to Whole Zn-finger Inactivated Virus Stimulation and Various HIV-1 Peptide Antigens
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 4 | 6
cells/mm^3
  HIV-1 MN | 0.6 [0 to 0.6] | 0.1 [0.1 to 0.2] | 0 [0 to 0.7] | 0 [0 to 0.1]
  gag/pol/env | 0.1 [0.1 to 0.3] | 0 [0 to 0.2] | 0 [0 to 0.1] | 0.1 [0 to 0.3]
  tat/rev | 0.2 [0 to 0.4] | 0 [0 to 0.1] | 0 [0 to 0] | 0.1 [0 to 0.4]
  SEB | 16.9 [10.6 to 17.6] | 13.6 [7.0 to 19.5] | 7.9 [5.0 to 11.5] | 12.7 [8.2 to 15.8]

24. Secondary Outcome: Time-averaged AUC of T-cell Percent of HIV-1-specific CD4+ T-cell Subsets, Based on Flow Cytometry to Detect Antigen-specific IL-2-producing Cells Responding to Whole Zn-finger Inactivated Virus Stimulation and Various HIV-1 Peptide Antigens
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 4 | 6
percent
  HIV-1 MN | 0.1 [0 to 0.1] | 0 [0 to 0] | 0 [0 to 0.1] | 0 [0 to 0]
  gag/pol/env | 0 [0 to 0.1] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  tat/rev | 0 [0 to 0.1] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0.1]
  SEB | 2.1 [1.9 to 2.2] | 1.9 [1.8 to 2.4] | 1.5 [1.1 to 1.8] | 2.1 [1.6 to 2.9]

25. Secondary Outcome: Time-averaged AUC of T-cell Count of HIV-1-specific CD8+ T-cell Subsets, Based on Flow Cytometry to Detect Antigen-specific IL-2-producing Cells Responding to Whole Zn-finger Inactivated Virus Stimulation and Various HIV-1 Peptide Antigens
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 5 | 4 | 6
cells/mm^3
  HIV-1 MN | 0 [0 to 0.3] | 0.1 [0.1 to 0.3] | 0 [0 to 1.3] | 0.1 [0 to 0.1]
  gag/pol/env | 0.3 [0 to 0.3] | 0.3 [0 to 0.5] | 0 [0 to 0.3] | 0 [0 to 0.1]
  tat/rev | 0.3 [0.1 to 0.5] | 0 [0 to 0.2] | 0 [0 to 0.1] | 0 [0 to 0.1]
  SEB | 1.9 [1.4 to 2.8] | 5.3 [3.4 to 9.2] | 4.2 [2.9 to 5.7] | 2.1 [1.1 to 3.5]

26. Secondary Outcome: Time-averaged AUC of T-cell Percent of HIV-1-specific CD8+ T-cell Subsets, Based on Flow Cytometry to Detect Antigen-specific IL-2-producing Cells Responding to Whole Zn-finger Inactivated Virus Stimulation and Various HIV-1 Peptide Antigens
Description: as for outcome 9
Time Frame: From start of study vaccination to week 24
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 5 | 6 | 4 | 6
percent
  HIV-1 MN | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0.2] | 0 [0 to 0]
  gag/pol/env | 0.1 [0 to 0.1] | 0 [0 to 0.1] | 0 [0 to 0] | 0 [0 to 0]
  tat/rev | 0 [0 to 0.1] | 0 [0 to 0.1] | 0 [0 to 0] | 0 [0 to 0]
  SEB | 0.3 [0.3 to 0.4] | 0.5 [0.3 to 1.5] | 0.7 [0.4 to 1.4] | 0.3 [0.2 to 0.5]

27. Secondary Outcome: Lymphocyte Proliferation Stimulation Index (SI) in Response to Whole HIV-1 Antigen, p24 Antigen, and Pooled HIV-1 Peptide Antigens
Description: The assay was not run due to published data showing that this assay is less sensitive than the PHPC assays (used in secondary outcomes 4 and 5). There are no data available for the analysis.
Time Frame: From start of study vaccination to week 24
Population: There are no data available for the analysis.
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

28. Other Pre Specified Outcome: Breadth of HIV-1-specific Immune Response, as Determined by the Number of Overlapping HIV-1 Peptides for Which the ELISPOT Assay for IFN-gamma Production is Observed to Have Five or More Spot-forming Cells/ 10^5 PBMCs
Description: Additional outcome measure for possible supportive exploratory analysis. The assay was not run due to published data showing that this assay is less sensitive than the PHPC assays (used in secondary outcomes 4 and 5). There are no data available for the analysis.
Time Frame: From start of study vaccination to week 24
Population: There are no data available for the analysis.
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study vaccination to week 61
Arm/Group | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 6/6 | 6/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A: 0.1 mg DNA/Participant Vaccination at Weeks 1, 7, 13 (N=6) | C: 0.4 mg DNA/Participant Vaccination at Weeks 1, 7, 13 (N=6) | E: 0.4 mg DNA/Participant Vaccination at Weeks 0,1,6,7,12,13 (N=6) | Placebo (N=7)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Lacrimation decreased (Eye disorders) | 0 | 1 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0 | 2
Injection site discomfort (General disorders) | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 3
Injection site mass (General disorders) | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1
Injection site pruritus (General disorders) | 3 | 0 | 1 | 1
Malaise (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Vaccination site erythema (General disorders) | 1 | 0 | 0 | 0
Vaccination site pain (General disorders) | 0 | 0 | 2 | 0
Vaccination site reaction (General disorders) | 1 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1
Secondary syphilis (Infections and infestations) | 1 | 0 | 0 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood bicarbonate (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Blood glucose abnormal (Investigations) | 1 | 1 | 1 | 0
Blood glucose decreased (Investigations) | 0 | 2 | 0 | 1
Blood phosphorus decreased (Investigations) | 2 | 1 | 1 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2 | 4 | 3
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0

LIMITATIONS AND CAVEATS:
This is a Phase I/II small sample study that was not powered for the secondary efficacy endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.